CLINICAL TRIAL: NCT07185594
Title: A Phase Ⅱ/Ⅲ Study to Evaluate the Efficacy and Safety of HRS-2129 for Postsurgical Pain Management in Abdominal Surgery
Brief Title: A Phase Ⅱ/Ⅲ Study of HRS-2129 for Postsurgical Pain Management in Abdominal Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-2129-301
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- HRS-2129 low-dose group (Experimental)
  Interventions: Drug: HRS-2129 Tablets; Drug: Blank Preparation.
- HRS-2129 middle-dose group (Experimental)
  Interventions: Drug: HRS-2129 Tablets; Drug: Blank Preparation.
- HRS-2129 high-dose group (Experimental)
  Interventions: Drug: HRS-2129 Tablets; Drug: Blank Preparation.
- Blank preparation placebo group (Placebo Comparator)
  Interventions: Drug: Blank Preparation.
- Tramadol Hydrochloride SR Tablets group (Active Comparator)
  Interventions: Drug: Tramadol Hydrochloride SR Tablets

INTERVENTIONS:
Drug: HRS-2129 Tablets — HRS-2129 tablets.
  Arms: HRS-2129 high-dose group; HRS-2129 low-dose group; HRS-2129 middle-dose group
Drug: Blank Preparation. — Blank preparation.
  Arms: Blank preparation placebo group; HRS-2129 high-dose group; HRS-2129 low-dose group; HRS-2129 middle-dose group
Drug: Tramadol Hydrochloride SR Tablets — Tramadol Hydrochloride SR tablets.
  Arms: Tramadol Hydrochloride SR Tablets group

SUMMARY:
This is a phase II/III, multi-center, randomized, double-blind, comparator-controlled study to evaluate the efficacy and safety of HRS-2129 for postoperative pain management in abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form before initiating trial-related activities, fully understand the purpose and significance of this trial, and voluntarily comply with the trial procedures;
2. Scheduled to undergo abdominal surgery (laparotomy or laparoscopy) under general anesthesia;
3. Aged ≥ 18 years (based on the date of signing the informed consent form), regardless of gender;
4. Body Mass Index (BMI) between 18.0 kg/m² and 30.0 kg/m² (inclusive);
5. American Society of Anesthesiologists (ASA) Physical Status Classification Grade I to II;
6. Within 6 hours after surgery (timed from the completion of the last suture), the subject has a Resting Pain Numeric Rating Scale (NRS) score ≥ 4 at any time point;
7. Male and female subjects of childbearing potential must agree to use effective contraceptive measures together with their partners from the time of signing the informed consent form until 1 month after the last administration of the investigational product, with no childbearing plans and no intention to donate sperm/eggs; Female subjects of childbearing potential must have a negative serum pregnancy test within 3 days before the first administration (or within 2 days before surgery) and must not be breastfeeding.

Exclusion Criteria:

1. Subjects with a history of asthma, chronic urticaria, severe allergic reactions (see Appendix 13.11 for details), allergies to multiple (3 or more) drugs or foods, as well as a personal history or family history of hereditary angioedema before randomization;
2. Subjects with a history of new-onset myocardial infarction or unstable angina pectoris within 6 months before randomization, or a history of New York Heart Association (NYHA) Heart Failure Classification Grade II or higher;
3. Subjects with a history of arrhythmia requiring treatment before surgery;
4. Subjects who developed severe arrhythmia during surgery and were deemed unsuitable for participation in this study by the investigator;
5. Subjects with a history of malignant tumor within 5 years before randomization (except for cutaneous squamous cell carcinoma or cutaneous basal cell carcinoma that has been completely resected and is clinically stable);
6. Subjects with a previous history of motion sickness, and the investigator judges that they may experience nausea and vomiting after surgery;
7. Subjects with a history of mental system diseases (such as schizophrenia, depression, etc.) and cognitive impairment before randomization;
8. Subjects with concurrent pain in various parts of the body, which the investigator believes may confuse the assessment of postoperative pain Subjects with a history of pheochromocytoma before randomization;
9. Subjects with concurrent conditions that the investigator believes may affect pain assessment, such as skin or neurological lesions in the affected skin area that may affect sensation;
10. Subjects with a previous surgical history at the surgical site;
11. QTc interval at screening: > 450 ms for males and > 470 ms for females (QTc calculated using the Fridericia formula); other electrocardiographic abnormalities that are clinically significant as judged by the investigator, which may affect the subject's safety or cause distress to the subject's participation in this clinical trial;
12. Subjects with hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg) or hypotension (systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg) at screening, excluding abnormalities occurring during the period from entry into the operating room to exit from the recovery room;
13. Subjects with laboratory test abnormalities at screening;
14. Positive hepatitis B surface antigen (HBsAg) or positive hepatitis C virus antibody (HCV Ab) at screening (further testing for hepatitis B virus deoxyribonucleic acid (HBV DNA) titer or hepatitis C virus ribonucleic acid (HCV RNA) is required; subjects with results exceeding the detection limit of the assay must be excluded); positive human immunodeficiency virus antibody (HIV Ab); positive serum treponema pallidum antibody (TP Ab) (further testing for treponema pallidum titer is required; subjects with positive results must be excluded);
15. Participation in any other clinical study within 3 months before randomization;
16. Use of other drugs that affect analgesic efficacy before screening, where the time from the last dose to randomization is less than 5 times the drug's half-life;
17. Other circumstances where the investigator judges that the subject is unsuitable for participation in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The time-weighted sum of differences in resting pain intensity within 48 hours after the start of administration of the investigational product. | Within 48 hours after the start of administration of the investigational product.

SECONDARY OUTCOMES:
The time-weighted sums of differences in resting pain intensity at 6 hours, 12 hours, 16 hours, 24 hours, within 12 hours-24 hours, and within 24 hours-48 hours after the start of administration (Sum of Pain Intensity Difference, SPID). | At 6 hours, 12 hours, 16 hours, 24 hours, within 12 hours-24 hours, and within 24 hours-48 hours after the start of administration.
The time-weighted sums of differences in movement-related pain intensity at 6 hours, 12 hours, 16 hours, 24 hours, within 12 hours-24 hours, and within 24 hours-48 hours after the start of administration. | At 6 hours, 12 hours, 16 hours, 24 hours, within 12 hours-24 hours, and within 24 hours-48 hours after the start of administration.
Proportion of subjects with a reduction of ≥30%, ≥50%, and ≥70% in resting pain Numeric Rating Scales (NRS) scores from baseline at 24 hours and 48 hours after the first dose. | At 24 hours and 48 hours after the first dose.
Proportion of subjects with a reduction of ≥30%, ≥50%, and ≥70% in movement-related pain NRS scores from baseline at 24 hours and 48 hours after the first dose. | At 24 hours and 48 hours after the first dose.
Percentage of subjects who did not use rescue analgesics within 0-24 hours, 24-48 hours, and 0-48 hours after the first dose. | Within 0-24 hours, 24-48 hours, and 0-48 hours after the first dose.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided